CLINICAL TRIAL: NCT04383548
Title: Randomized Prospective Clinical Study for Efficacy of Anti-Corona VS2 Immunoglobulins Prepared From COVID19 Convalescent Plasma in Prevention of Infection in High Risk Groups as Well as Treatment of Early Cases of COVID19 Patients
Brief Title: Clinical Study for Efficacy of Anti-Corona VS2 Immunoglobulins Prepared From COVID19 Convalescent Plasma Prepared by VIPS Mini-Pool IVIG Medical Devices in Prevention of SARS-CoV-2 Infection in High Risk Groups as Well as Treatment of Early Cases of COVID19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshaimaa Mokhtar Selim mohamed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mini-pooled IVIG in COVID19
Record Dates: First submitted 2020-04-17; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyper immunoglobulins have anti-Corona VS2 immunoglobulin (Experimental): safe purified hyper immunoglobulins containing anti-Corona VS2 immunoglobulins from plasma collected from COVID19 convalescent patients
  Interventions: Other: hyper immunoglobulins containing anti-Corona VS2 immunoglobulin

INTERVENTIONS:
Other: hyper immunoglobulins containing anti-Corona VS2 immunoglobulin — Prospective randomized clinical study for efficacy of anti-SARS-CoV-2 hyper immunoglobulins prepared from COVID19 convalescent plasma using VIPS Mini-Pool IVIG medical device

SUMMARY:
Preparation of safe purified hyper immunoglobulins containing anti-Corona VS2 immunoglobulins from plasma collected from COVID19 convalescent patients to be used to:

1. To determine efficacy of COVID19 hyper immunoglobulins prepared from convalescent plasma using VIPS Mini-Pool IVIG medical device in the treatment of COVID19
2. To determine efficacy of anti-SARS-CoV-2 hyper immunoglobulins in the prevention of infection in high risk groups exposed to SARS-CoV-2 infection

DETAILED DESCRIPTION:
The current COVID19 pandemic poses a huge challenge on health authorities and infrastructure due to rapid progression of infection with an estimated rate of severe disease that needs hospitalization and medical intervention. It is also noteworthy that health care workers are at high risk of contracting COVID19 when dealing with cases.

Previous experience with Corona SARS demonstrated a therapeutic benefit of using convalescent plasma for patients with Corona SARS in Hong Kong. Passive immunization using hyper immunoglobulin preparations against measles as well as early treatment was proven effective when compared to no intervention conservative approach . A recent publication encourages the use of COVID19 convalescent serum for the preparation of hyper immunoglobulins to be used for passive immunization as well as treatment of early disease before the development of lower respiratory tract disease; pneumonia.

Provision of Convalescent COVID19 hyper immunoglobulin:

This can be achieved through one of the following three approaches:

Fist approach: Convalescent COVID19 immunoglobulins can be obtained by transfusion of 1 - 4 units of COVID19 FFP for passive immunization or treatment of early disease. The advantages of this approach is that it is easy to prepare such units of FFP through regular blood banks. Disadvantages include variability of existence and levels of neutralizing COVID19 immunoglobulins in individual plasma units. This may result in variability of effectiveness for such an approach for prevention and treatment. Risk of transfusion transmitted infections as well as immunological adverse events due to infusion of large volume of FFP are among other disadvantages of using individual FFP units.

Second approach: Classical industrial COVID19 hyper immunoglobulins from convalescent donors. This approach provides more consistent small volumes of concentrated hyperimmunoglobulin preparations due to pooling of plasma donations from large number of convalescent donors which bypasses the variability of neutralizing immunoglobulins in individual plasma donations. The preparation of hyper immunoglobulins includes steps for virus inactivation which results in safer products compared to non-virally inactivated FFP. Production of COVID19 convalescent hyper immunoglobulins under current situation is practically not feasible due to limited source COVID19 convalescent plasma, regulatory hurdles and the large volume of production batches (minimum of 100s of liters of convalescent plasma).

Third approach: Recently a Swiss company developed medical device to prepare Intravenous Immunoglobulin (IVIG) preparations from only 4 liters of plasma (20 units of FFP) which is sufficient to produce 20 grams of IVIG. The technology involves the concentration of immunoglobulins from 20 plasma donations into IVIG preparations as well as virus inactivation of lipid enveloped viruses (HBV, HCV, HIV & Corona VS2) . Safety of Mini-Pool IVIG was proven in a previous clinical trial conducted in ITP pediatric population. The yield of one batch of this Mini-Pool IVIG is about 20 gms which can be sufficient for prophylaxis and/or treatment of 6 - 10 individuals.

ELIGIBILITY:
Inclusion Criteria:

a. Passive immunization group (Group A)

1. 20 high risk exposed persons (HCPs) who are nasopharyngeal swab SARSCoV-2 PCR negative and seronegative for SARS-CoV-2 IgM/IgG antibodies to receive prophylactic anti- SARS-CoV-2 hyper immunoglobulin. Selected population can be both male and female with age range 21 - 50 years b. 20 high risk persons (HCPs) who are nasopharyngeal swab SARS-CoV-2 PCR negative and seronegative for SARS-CoV-2 IgM/IgG antibodies as control group. Selected population can be both male and female with age range 21 - 50 years
2. Patient group (group B):

a. 30 patients with COVID19 disease and nasopharyngeal swab or sputum SARSCoV-2 positive PCR to receive anti-SARS-CoV-2 in addition to applied clinical management protocol. Selected test group can be male or female with age >20 years b. 30 patients with COVID-19 disease and nasopharyngeal swab or sputum SARS-CoV-2 PCR positive managed according to applied clinical management protocols of COVID-19 disease as control group. Selected test group can be male or female with age >30 years

Exclusion Criteria:

1. Passive immunization group (Group A):

   1. Age less than 21 or above 50 years
   2. . Nasopharyngeal swab SARS-CoV-2 positive PCR
   3. . Presence of anti-SARS-CoV-2 IgM, IgG
   4. Presence of comorbidities such as hypertension, diabetes, chronic renal disease, previous thrombotic events or states of allergy such as urticaria or bronchial asthma as well as previous adverse events due to infusion of IVIG
2. Patient group (group B):

   1. Age less than 20 years
   2. . SARS-CoV-2 PCR negative
   3. . COVID-19 patients who may suffer from co morbidities such as hypertension, diabetes, chronic renal disease, thrombotic tendency or history of adverse events to IVIG as well as old age will be excluded to reduce the possibility of development of serious adverse events related to infusion of IVIG unless it will be for compassionate use in advanced stages of COVID-19 patients and after obtaining informed consent

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of COVID19 hyper immunoglobulins for patients | 2 weeks
  efficacy of COVID19 hyper immunoglobulins prepared from convalescent plasma using VIPS Mini-Pool IVIG medical device in the treatment of COVID19
Efficacy of COVID19 hyper immunoglobulins for high risk groups | 1 month
  efficacy of anti-SARS-CoV-2 hyper immunoglobulins in the prevention of infection in high risk groups exposed to SARS-CoV-2 infection
Safety of anti-SARS-CoV-2 hyper immunoglobulins assessed by percentage of adverse events | 72 hours
  overall percentage of adverse events as hemolysis and anaphylaxis ,headache and other complains that occur during 72 hours of following infusion of anti-SARS-CoV-2 hyper immunoglobulins will be assessed by 1-vital sign 2-hemolysis by LDH and bilirubin level

CONTACTS AND LOCATIONS:
Overall Officials: Maha A Mohamed, professor, Study Director — Assiut univeristy; Magdy El Ekiaby, Doctor, Principal Investigator — Sabrawishy hospital,Dokki,Giza,Egypt; Azza M Ez-Eldin, professor, Principal Investigator — Assiut univeristy; Alia M Hussein, professor, Principal Investigator — Assiut univeristy

REFERENCES:
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] El-Ekiaby M, Sayed MA, Caron C, Burnouf S, El-Sharkawy N, Goubran H, Radosevich M, Goudemand J, Blum D, de Melo L, Soulie V, Adam J, Burnouf T. Solvent-detergent filtered (S/D-F) fresh frozen plasma and cryoprecipitate minipools prepared in a newly designed integral disposable processing bag system. Transfus Med. 2010 Feb;20(1):48-61. doi: 10.1111/j.1365-3148.2009.00963.x. Epub 2009 Sep 23. PMID 19778318